CLINICAL TRIAL: NCT01037790
Title: Phase II Trial of the Cyclin-Dependent Kinase Inhibitor PD 0332991 in Patients With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03909
Record Dates: First submitted 2009-12-10; First posted 2009-12-23 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Adult Solid Tumor; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Adult Central Nervous System Germ Cell Tumor; Adult Teratoma; Benign Teratoma; Estrogen Receptor-negative Breast Cancer; Estrogen Receptor-positive Breast Cancer; Familial Testicular Germ Cell Tumor; HER2-negative Breast Cancer; HER2-positive Breast Cancer; Male Breast Cancer; Ovarian Immature Teratoma; Ovarian Mature Teratoma; Ovarian Monodermal and Highly Specialized Teratoma; Progesterone Receptor-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Recurrent Colon Cancer; Recurrent Extragonadal Germ Cell Tumor; Recurrent Extragonadal Non-seminomatous Germ Cell Tumor; Recurrent Extragonadal Seminoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Melanoma; Recurrent Ovarian Germ Cell Tumor; Recurrent Rectal Cancer; Stage III Extragonadal Non-seminomatous Germ Cell Tumor; Stage III Extragonadal Seminoma; Stage III Malignant Testicular Germ Cell Tumor; Stage III Ovarian Germ Cell Tumor; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Extragonadal Non-seminomatous Germ Cell Tumor; Stage IV Extragonadal Seminoma; Stage IV Melanoma; Stage IV Ovarian Germ Cell Tumor; Stage IV Rectal Cancer; Testicular Immature Teratoma; Testicular Mature Teratoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Teratoma; Breast Neoplasms, Male; Breast Neoplasms; Testicular Neoplasms; Melanoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 - Metastatic breast cancer (Experimental): Metastatic breast cancer
  PD-0332991 Given orally, 125 mg QD on a 21-day
  Interventions: Drug: PD-0332991
- Arm 2 - Metastatic colorectal cancer that harbors the Kras or BRAF mutation (Experimental): Metastatic colorectal cancer that harbors the Kras or BRAF mutation
  PD-0332991 Given orally, 125 mg QD on a 21-day
  Interventions: Drug: PD-0332991
- Arm 3 - Advanced or metastatic esophageal and/or gastric cancer (Experimental): Advanced or metastatic esophageal and/or gastric cancer
  PD-0332991 Given orally, 125 mg QD on a 21-day
  Interventions: Drug: PD-0332991
- Arm 4 - Cisplatin-refractory, unresectable germ cell tumors (Experimental): Cisplatin-refractory, unresectable germ cell tumors
  PD-0332991 Given orally, 125 mg QD on a 21-day
  Interventions: Drug: PD-0332991
- Arm 5 - CCND1amplification, CDK4/6mutation, CCND2amplification, OR other functional G1/S alterations (Experimental): Any tumor type if tissue tests positive for CCND1 amplification, CDK4/6 mutation , CCND2 amplification OR any other functional alteration at the G1/S checkpoint.
  PD-0332991 Given orally, 125 mg QD on a 21-day
  Interventions: Drug: PD-0332991

INTERVENTIONS:
Drug: PD-0332991 — Given orally, 125 mg QD on a 21-day
  Other Names: Palbociclib

SUMMARY:
RATIONALE: PD 0332991 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects and how well PD 0332991 works in treating patients with refractory solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rates following treatment with PD 0332991 in the following malignancies: 1) Metastatic breast cancer, 2) Metastatic colorectal cancer, 3) Metastatic melanoma with CDK4 mutation or amplification, or 4) Cisplatin-refractory, unresectable germ cell tumors.

OUTLINE:

Patients receive oral PD 0332991 once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

- Disease Characteristics:

All Subjects: All subjects treated under this protocol will have histologically documented cancer of one of the following types:

A. Metastatic breast cancer (7 triple negative, 23 ER+ after the first 15 patients are enrolled on the non-CCND1cohort; in addition 10 HER2+ for combination trastuzumab and PD0332991 therapy) up to 55 total enrollment slots B. Metastatic colorectal cancer that harbors the Kras or BRAF mutation (15-30 enrollment slots) C. Advanced or metastatic esophageal and/or gastric cancer (15-30 enrollment slots) D. Cisplatin-refractory, unresectable germ cell tumors (15-30 enrollment slots) E. Any tumor type if tissue tests positive for CCND1 amplification, CDK4/6 mutation, CCND2 amplification OR any other functional alteration at the G1/S checkpoint. (15-30 enrollment slots)

- Biopsy Requirements: For Subjects with accessible disease amenable to biopsy: A biopsy will be obtained pre-treatment and in during cycle 1 (while patient is receiving drug) for molecular markers of the cell cycle, and its inhibition.

* Subjects will be > 18 years old
* The subject has disease that is assessable by tumor marker, physical, or radiologic means.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The subject has adequate organ function, defined as follows A. Bilirubin ≤ 1.5 x the upper limit of normal (ULN) B. Serum creatinine ≤ 1.5 x UNL or calculated creatinine clearance ≥ 60 mL/min, and C. For subjects without liver metastases: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN D. For subjects with liver metastases: alanine aminotransferase (ALT) and aspartate aminotransferase ≤ 5 x ULN
* All tumors must test positive for Rb expression except:

A. ER positive metastatic breast tumors (data now shows all to be Rb positive.) B. Any tumor type if tissue tests positive for CCND1 amplification, CDK4/6 mutation, CCND2 amplification OR any other functional alteration at the G1/S checkpoint.

- The subject has adequate marrow function, defined as follows: A. Absolute neutrophil count (ANC) >1500/mm3 B. Platelets >100,000/mm3, and C. Hemoglobin > 9 g/dL

* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Sexually active subjects (male and female) must use accepted methods of contraception during the course of the study and for 3 months after the last dose of protocol drug(s).
* Female subjects of childbearing potential must have a negative pregnancy test at screening. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months.
* However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, or ovarian suppression.

Exclusion Criteria

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) within 3 weeks (or nitrosoureas or mitomycin C within 6 weeks) before the first dose of PD 0332991. . Patients with HER2-overexpressing tumors may receive trastuzumab up to the date of starting therapy, and may continue to receive trastuzumab while receiving PD0332991.
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* The subject has not recovered from clinically-meaningful toxicity due to prior therapy (i.e., back to baseline or Grade ≤ 1), with the exception of neurotoxicity and alopecia.
* The subject has untreated or uncontrolled brain metastases or evidence of leptomeningeal involvement of disease unless the subject has a teratoma in which case s/he may be eligible if all other eligibility criteria are met
* The subject has uncontrolled intercurrent illness including, but not limited to:

  1. ongoing or active infection
  2. diabetes mellitus
  3. hypertension
  4. symptomatic congestive heart failure, unstable angina pectoris, stroke or myocardial infarction within 3 months
* The subject has a baseline corrected QT interval (QTc) > 470 ms.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV). Note:

baseline HIV screening is not required

- The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter ODwyer, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Karasic TB, O'Hara MH, Teitelbaum UR, Damjanov N, Giantonio BJ, d'Entremont TS, Gallagher M, Zhang PJ, O'Dwyer PJ. Phase II Trial of Palbociclib in Patients with Advanced Esophageal or Gastric Cancer. Oncologist. 2020 Dec;25(12):e1864-e1868. doi: 10.1634/theoncologist.2020-0681. Epub 2020 Aug 8. PMID 32692450
- [Derived] McAndrew NP, Dickson MA, Clark AS, Troxel AB, O'Hara MH, Colameco C, Gallager M, Gramlich K, Zafman K, Vaughn D, Schwartz GK, O'Dwyer PJ, DeMichele A. Early treatment-related neutropenia predicts response to palbociclib. Br J Cancer. 2020 Sep;123(6):912-918. doi: 10.1038/s41416-020-0967-7. Epub 2020 Jul 9. PMID 32641862

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Metastatic breast cancer
  PD-0332991: Given orally, 125 mg QD on a 21-day
- Arm 2: Metastatic colorectal cancer that harbors the Kras or BRAF mutation
  PD-0332991: Given orally, 125 mg QD on a 21-day
- Arm 3: Advanced or metastatic esophageal and/or gastric cancer
  PD-0332991: Given orally, 125 mg QD on a 21-day
- Arm 4: Cisplatin-refractory, unresectable germ cell tumors
  PD-0332991: Given orally, 125 mg QD on a 21-day
- Arm 5: Any tumor type if tissue tests positive for CCND1 amplification, CDK4/6 mutation , CCND2 amplification OR any other functional alteration at the G1/S checkpoint.
  PD-0332991: Given orally, 125 mg QD on a 21-day
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
Started | 63 | 18 | 19 | 30 | 11
Completed | 63 | 18 | 19 | 30 | 11
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Total
Number analyzed (Participants) | 63 | 18 | 19 | 30 | 11 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 48 | 10 | 11 | 29 | 11 | 109
  >=65 years | 15 | 8 | 8 | 0 | 0 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 8 | 4 | 4 | 9 | 88
  Male | 0 | 10 | 15 | 26 | 2 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black | 3 | 1 | 1 | 3 | 0 | 8
  Other | 2 | 1 | 0 | 4 | 0 | 7
  White | 58 | 16 | 18 | 23 | 11 | 126
Region of Enrollment [Number; unit: participants]
  United States | 63 | 18 | 19 | 30 | 11 | 141

OUTCOME MEASURES:

1. Primary Outcome: Response Rates
Description: Response rates will be measured using the Response Evaluation Criteria in Solid Tumors (RECIST):
  Complete Response (CR) - Disappearance of all target lesions Partial Response (PR) - ≥30% decrease in the sum of the longest diameter of the target lesions compared with baseline Progressive Disease (PD) - ≥20% increase in the sum of the longest diameter of the target lesions compared with the smallest sum of the longest diameter recorded since treatment started OR The appearance of 1 or more new lesions Stable Disease (SD) - Neither PR or PD Not Evaluable (NE)
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
Number analyzed (Participants) | 63 | 18 | 19 | 30 | 11
Participants
  partial response | 4 | 0 | 0 | 0 | 0
  stable disease | 32 | 6 | 6 | 17 | 3
  progressive disease | 25 | 8 | 4 | 9 | 7
  not evaluable for response | 2 | 4 | 9 | 4 | 1

ADVERSE EVENTS:
Time Frame: 10years
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/18 | 1/19 | 0/30 | 1/11
Serious Adverse Events (participants affected / at risk) | 1/63 | 10/18 | 11/19 | 10/30 | 4/11
Other Adverse Events (participants affected / at risk) | 40/63 | 18/18 | 19/19 | 25/30 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=63) | Arm 2 (N=18) | Arm 3 (N=19) | Arm 4 (N=30) | Arm 5 (N=11)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
elevated alk phos (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
elavated ALT (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
elevated AST (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GI bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
leukopenia (Investigations) | 0 (0) | 5 (5) | 4 (4) | 10 (10) | 0 (0)
lymphopenia (Investigations) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
neutropenia (Investigations) | 0 (0) | 6 (6) | 6 (6) | 10 (10) | 2 (2)
thrombocytopenia (Investigations) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 2 (2)
thromboembolic event (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=63) | Arm 2 (N=18) | Arm 3 (N=19) | Arm 4 (N=30) | Arm 5 (N=11)
aches (General disorders) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 34 (34) | 10 (10) | 7 (7) | 7 (7) | 5 (5)
anorexia (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 5 (5) | 3 (3) | 0 (0)
arthalgia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
belching (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
blurred vision (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bruising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
burning eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 13 (13) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
dry eyes (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dysguesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
early satiety (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
elevated alk phos (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
elavated ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
elevated AST (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
elevated creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 28 (28) | 8 (8) | 9 (9) | 9 (9) | 2 (2)
fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
flu (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GI bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
heartburn (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hiccups (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
hyperbilirubinemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
joint stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
leukopenia (Investigations) | 17 (17) | 0 (0) | 9 (9) | 11 (11) | 2 (2)
lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
liver pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lower extemity edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lymphopenia (Investigations) | 10 (10) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
mouth sensitivity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
mucositis (Gastrointestinal disorders) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
myalgia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nausea (Nervous system disorders) | 9 (9) | 7 (7) | 4 (4) | 4 (4) | 2 (2)
neck pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
neutropenia (Investigations) | 18 (18) | 6 (6) | 7 (7) | 9 (9) | 1 (1)
night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nipple sensitivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
orthostasis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
seasonal allergies (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
sinus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
thrombocytopenia (Investigations) | 26 (26) | 10 (10) | 9 (9) | 9 (9) | 6 (6)
thromboembolic event (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
unsteady gait (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (3) | 2 (2)
weight loss (Investigations) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT01037790/Prot_000.pdf